CLINICAL TRIAL: NCT06570018
Title: Short Term Outcome Following Post Operative Enhanced Recovery Implementation in Patients With Perforated Peptic Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amna A. Desouky, MD, Assisstant professor of Medical Surgical Nursing, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Enhanced recovery
Record Dates: First submitted 2024-08-20; First posted 2024-08-26 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Emergent Surgery; Perforated Peptic Ulcer
MeSH Terms: conditions — Peptic Ulcer Perforation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced recovery group (Experimental): who received postoperative enhanced recovery after open surgical repair for perforated peptic ulcer
  Interventions: Procedure: Post operative enhanced recovery elements
- Control group (No Intervention): who exposed to standard care

INTERVENTIONS:
Procedure: Post operative enhanced recovery elements — According to the study group the researchers collaborated with surgeons, nurses, and anesthesiologists to implement post operative enhanced recovery protocol that defined clearly in the following elements Early nutrition, Early mobilization, Non-opioid analgesia. Early removal of abdominal drains and tubes throughout the patients' hospital stay up to their discharge.
  Arms: Enhanced recovery group

SUMMARY:
This study aimed to evaluate the effect of implementing post operative enhanced recovery on perforated peptic ulcer surgery outcome.

The current study anticipated better outcomes in the form of early functional recovery, reduced length of hospital stays, less thirty days post operative morbidity, and better gastrointestinal quality of life after implementing post operative enhanced recovery in patients with perforated peptic ulcer.

DETAILED DESCRIPTION:
This study aimed to evaluate the effect of implementing post operative enhanced recovery on perforated peptic ulcer surgery outcomes.

Methods: Quasi- experimental research design was utilized. The study was conducted at Assiut University Hospital.

A purposive sample of thirty patients (study group) who received postoperative enhanced recovery after open surgical repair of perforated peptic ulcer compared with thirty patients (control group) who exposed to routine care.

patient assessment sheet and gastrointestinal quality of life index were the tools used for data collection.

ELIGIBILITY:
Inclusion Criteria:

* Age ranged from 18 to 65 years,
* Diagnosed with perforated peptic ulcer,
* Ulcer size less than 10 mm.
* Underwent emergent surgical intervention

Exclusion Criteria:

* Malignant ulcer.
* Other GIT diseases (corn's disease & ulcerative colitis)
* Pregnant women
* Psychiatric or neurological illness.
* Who refused to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal functional recovery (first bowel movement) | Within the first 24 hours postoperative or more
  Tool; Patient assessment sheet
  * It was developed by researchers based on literatures review to assess postoperative clinical data (part 2) as gastrointestinal functional recovery (first bowel movement) through physical examination.
  * The mean score of time for two groups was compared
Gastrointestinal functional recovery(first flatus passage) | Within the first 24 hours postoperative or more
  Tool; Patient assessment sheet
  * It was developed by researchers based on literatures review to assess postoperative clinical data (part 2) as gastrointestinal functional recovery (first flatus passage) through physical examination.
  the mean score of time for two groups was compared
Gastrointestinal functional recovery(first stool passage) | First stool passage within three days postoperative or more
  Tool; Patient assessment sheet
  - It was developed by researchers based on literatures review to assess postoperative clinical data (part 2) as gastrointestinal functional recovery (first stool passage) postoperative.through health history.
  The mean score of time for two groups was compared
postoperative complications | Immediately post operative up to thirty days postoperative
  post operative complications included complications that occured within 30- days post operative. Every patient had been assessed for developing pneumonia, admission to critical care, abdominal collection, intra-abdominal abscess, suture leakage, omental patch leakage, septic shock, prolonged ileus, surgical site infection, urinary tract infection, deep venous thrombosis (DVT), and reoperation
Legnth of hospital stay | seven days up to two weeks
  Hospitalization duration from admission up to discharge Mean score of days for two groups will be compared.

SECONDARY OUTCOMES:
gastrointestinal quality of life | Before hospital dicharge and after thirty days postoperative
  gastrointestinal quality of life was evaluated for all patients before discharge and after thirty days postoperative using Gastrointestinal quality of life index (Eypasch, 1993).
  It is a 36-item scale divided into five domains; GIT symptoms (10 items), physical (6 items), emotion (6 items), social (2 items) and disease specific (8 items) Cronbach's alpha was 0.89
  Scoring:
  Each item is based on a 0-4 Likert scale with 0 being least desirable to 4 being the most desirable option. The total scores represent Gastrointestinal Quality of Life Index. It ranges from 0 to 144 with higher scores indicating a better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Ayoub, Ass. prof., Principal Investigator — Assiut University -Assiut city
Locations (1):
- Faculty of Nursing, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Desoky AA, Ayoub MT, Mostafa NM, Hashem EM, Mohammed MA. Short-term outcome following postoperative enhanced recovery implementation in patients with perforated peptic ulcer. Eur J Med Res. 2025 Apr 4;30(1):234. doi: 10.1186/s40001-025-02432-7. PMID 40186297